CLINICAL TRIAL: NCT04110743
Title: EXPLORER PET/CT: A Pilot Evaluation in Healthy Volunteers
Brief Title: EXPLORER PET/CT in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1341792
Record Dates: First submitted 2019-09-18; First posted 2019-10-01 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2023-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- delayed imaging acquisition (Other): 10 mCi of 18F fluorodeoxyglucose (FDG) will be injected through the IV and a 60-minute dynamic scan will begin on EXPLORER. The IV line will be removed after dynamic acquisition. The dynamic scan will be preceded by ultra low-dose (1.298 mSv) CT scan to provide information for attenuation correction for the PET data. At 90 minutes, 3-, 6-, 9- and 12-hours, a static whole-body scan for 20 minutes will be acquired on EXPLORER. Prior to the 90-minute scan a low-dose CT (7.44 mSv) will be obtained both for anatomic localization and for attenuation correction purposes. Prior to each of the later time-points (3-, 6-, 9- and 12-hours), an ultra low-dose (1.298 mSv) CT scan will be acquired. This scan will be for attenuation correction purposes only. Following the 12-hour scan, the participant's study visit will be completed. MRI Brain will be also obtained after PET/CT scanning for anatomic correlation.
  Interventions: Device: EXPLORER PET/CT
- low FDG dose imaging (Other): 0.5 mCi of 18F-FDG (1/20th of the standard dose) will be hand injected through the IV and a 60-minute dynamic scan will begin on EXPLORER. The dynamic scan will be preceded by an ultra-low-dose CT scan (1.298 mSv) for attenuation correction. The standard 20-minute EXPLORER scan obtained at 90 minutes will be obtained after a low dose CT (7.44 mSv) for attenuation and co-localization. The standard 20-minute EXPLORER scan obtained at 3 hours will be preceded by an ultra-low-dose CT scan (1.298 mSv) for attenuation correction only. MRI Brain will be also obtained after PET/CT scanning for anatomic correlation.
  Interventions: Device: EXPLORER PET/CT
- comparison PET images reconstructed using CT-based attenuation (Other): 10 mCi of 18F-FDG will be hand injected through the IV and a 60-minute dynamic scan will begin on EXPLORER. Prior to the dynamic scan, an ultra-low-dose CT scan (1.298 mSv) will be acquired for attenuation correction purposes only. At 90 mins, a low dose non contrast enhancement CT (7.44 mSv) will be acquired vertex to toes. Iodinated contrast (150 cc of iodine Omnipaque 350) will then be intravenously injected (through the same IV placed to inject FDG) at 3 ml/sec while the patient remains still on the scanner and a second low-dose CT will be acquired. Finally, a 20-minute PET acquisition will be performed. The IV line will be removed after completion of the study. MRI Brain will be also obtained after PET/CT scanning for anatomic correlation.
  Interventions: Device: EXPLORER PET/CT

INTERVENTIONS:
Device: EXPLORER PET/CT — Intervention: PET/CT using different protocols

SUMMARY:
The objective of this pilot study is to collect preliminary data using total body scans on a new, first of its kind, FDA 510k-cleared positron emission tomography/computed tomography (PET/CT) scanner, called EXPLORER.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18 years of age or older
* Willing and able to fast for at least 6 hours before and for the duration of the scan
* Willing and able to lay motionless in a supine position for 60 and 20 minutes at separate timepoints.
* Willing and able to give informed consent

Exclusion Criteria:

* No Primary Care Physician
* Body weight >240 kg
* Allergy to iodine contrast (only for subjects enrolled in Arm 3)
* Creatinine levels > 1.5 mg/dL or estimated glomerular filtration rate (eGFR) < 60 ml/minute (only for subjects enrolled in Arm 3)
* Recent (1 month) contrast enhanced CT
* Any known concomitant acute infection (including upper respiratory infection, genitourinary infections, etc.
* History of metastatic or newly (last 5 years) diagnosed locally invasive cancer.
* Chemotherapy in the last 5 years
* Radiation therapy in the last 3 years
* Major surgery within the last 6 months.
* Pregnancy or breast-feeding
* Diabetes
* Fasting blood glucose level > 160 mg/dL before administration of FDG
* Prisoners
* The standard MRI contraindications apply, including but not limited to:

Having a pacemaker or other implanted electronic device. Metal foreign bodies, aneurysm clips, heart valve prosthesis, vascular stents, cochlear implants, embolization coils, gunshot wounds with retained bullet fragments, penile implant, IUCD.

Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Nardo, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Delayed Imaging Acquisition | Low FDG Dose Imaging | Comparison PET Images Reconstructed Using CT-based Attenuation
Started | 15 | 15 | 0
Completed | 15 | 15 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Arm 3 was not completed
Groups:
- Total: Total of all reporting groups
Arm/Group | Delayed Imaging Acquisition | Low FDG Dose Imaging | Comparison PET Images Reconstructed Using CT-based Attenuation | Total
Number analyzed (Participants) | 15 | 15 | 0 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  | 0
  Between 18 and 65 years | 14 | 15 |  | 29
  >=65 years | 1 | 0 |  | 1
Age, Continuous [Geometric Mean (Full Range); unit: YEARS] | 49.5 [26.1 to 78.6] | 45.3 [26.3 to 62.2] |  | 47.4 [26.1 to 78.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 |  | 16
  Male | 6 | 8 |  | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 |  | 0
  Not Hispanic or Latino | 0 | 0 |  | 0
  Unknown or Not Reported | 15 | 15 |  | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 0 | 1 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 0 | 0 |  | 0
  White | 7 | 10 |  | 17
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 8 | 4 |  | 12
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 |  | 30

OUTCOME MEASURES:

1. Primary Outcome: Standardized Uptake Value SUV(t)= C(t)/ID/BW; C(t) is Radioactivity Measured at the Time t, Decay Corrected to t=0 and Converted From a Volume to a Mass Based Unit Via the Factor 1/(1 g/mL); ID: the Injected Dose at t=0; W= Body Weight; SUV is Correct UM
Description: To collect preliminary data regarding FDG biodistribution in the organs listed as a function of time of 12 hours. Time-activity curves will be created
Time Frame: approximatively 12 hours for Arm 1 only
Measure: Mean (Standard Deviation); unit: SUV
Arm/Group | Delayed Imaging Acquisition
Number analyzed (Participants) | 15
SUV
  Aorta | 0.83 (0.47)
  Lungs | 0.48 (0.44)
  Liver | 1.68 (0.51)
  Spleen | 2.01 (0.49)
  Kidneys | 1.91 (0.83)
  Bone Marrow | 3.44 (0.85)
  Skeletal Muscles | 1.23 (0.44)
  Subcutaneous Fat | 0.25 (0.21)
  Whole Brain | 5.81 (1.87)
  Myocardium | 14.0 (6.93)

2. Primary Outcome: Coefficient of Variation. SD/Mean (Standard Deviation Divided by Mean Value)
Description: To obtain preliminary data regarding low dose EXPLORER noise level
Time Frame: approximatively 6 hours for Arm 1 only
Measure: Mean (Standard Deviation); unit: coefficient
Arm/Group | Delayed Imaging Acquisition
Number analyzed (Participants) | 15
coefficient
  Aorta | 60.5 (14.8)
  Lungs | 140.1 (8.1)
  Liver | 32.2 (9.0)
  Spleen | 31.4 (9.3)
  Kidneys | 64.4 (18.4)
  Bone Marrow | 40.8 (11.8)
  Skeletal Muscles | 53.0 (18.8)
  Subcutaneous Fat | 88.6 (24.8)
  Whole Brain | 54.5 (8.1)
  Myocardium | 63.0 (16.7)

3. Primary Outcome: Standardized Uptake Value
Description: To collect preliminary data about total body FDG perfusion and early biodistribution. Time-activity curves will be created
Time Frame: approximatively 90 minutes
Measure: Mean (Standard Deviation); unit: SUV
Groups:
- Arm 2: Average SUV mean at 90 minutes
Arm/Group | Delayed Imaging Acquisition | Arm 2
Number analyzed (Participants) | 15 | 15
SUV
  Aorta | 1.75 (0.34) | 0.88 (0.17)
  Lungs | 0.62 (0.37) | 0.32 (0.06)
  Liver | 2.49 (0.44) | 1.02 (0.19)
  Spleen | 2.15 (0.40) | 0.83 (0.15)
  Kidneys | 3.65 (1.85) | 1.45 (0.23)
  Bone Marrow | 2.51 (0.44) | 0.73 (0.15)
  Skeletal Muscles | 0.70 (0.19) | 0.37 (0.06)
  Subcutaneous Fat | 0.19 (0.05) | 0.19 (0.04)
  Whole Brain | 9.88 (2.63) | 4.95 (1.36)
  Myocardium | 10.73 (4.92) | 1.20 (0.80)

4. Primary Outcome: Standardized Uptake Value SUV(t)= C(t)/(ID/BW); C(t) is Radioactivity Measured From at Time t, Decay Corrected to t=0-converted From a Volume to a Mass Based Unit Via the Factor 1/(1 g/mL); ID: the Injected Dose at t=0; BW= Body Weight; SUV is Correct UM
Description: To obtain preliminary data to understand whether intravenous iodinated contrast agent produce a significant change in quantification of FDG uptake levels.
  Time/activity curves will be generated.
Time Frame: approximatively 3 hours
Measure: Mean (Standard Deviation); unit: SUV
Groups:
- Arm 2: average SUV mean obtained at 3 hours for Arm 2
Arm/Group | Delayed Imaging Acquisition | Arm 2
Number analyzed (Participants) | 15 | 15
SUV
  Aorta | 1.18 (0.30) | 0.39 (0.08)
  Lungs | 0.52 (0.53) | 0.15 (0.04)
  Liver | 2.11 (0.42) | 0.50 (0.10)
  Spleen | 2.09 (0.41) | 0.43 (0.08)
  Kidneys | 3.30 (1.34) | 0.66 (0.12)
  Bone Marrow | 2.92 (0.56) | 0.44 (0.09)
  Skeletal Muscles | 0.82 (0.21) | 0.21 (0.04)
  Subcutaneous Fat | 0.16 (0.05) | 0.07 (0.02)
  Whole Brain | 10.39 (3.02) | 2.97 (0.86)
  Myocardium | 11.60 (5.92) | 0.68 (0.59)

ADVERSE EVENTS:
Time Frame: AEs were collected during the study protocol activity of the one appointment for approximately 3 hours at which time the subject was off study.
Description: All participants were monitored for AEs and SAEs throughout their participation.
Arm/Group | Delayed Imaging Acquisition | Low FDG Dose Imaging | Comparison PET Images Reconstructed Using CT-based Attenuation
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/0
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/0

LIMITATIONS AND CAVEATS:
Logistical limitations did not allow us to enroll in Arm 3. It was originally expected that a CT with contrast could be completed on the EXPLORER scanner. It was learned during study activation that it could not. an additional limitation was finding research staff to complete follow up data collection delaying in reporting of the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/43/NCT04110743/Prot_SAP_000.pdf